CLINICAL TRIAL: NCT04706793
Title: A Phase 3, Double-Blind, Placebo-Controlled, 40-Week Extension Study to Assess the Efficacy and Safety of Etrasimod in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Oral Etrasimod Versus Placebo for the Treatment of Moderately to Severely Active Ulcerative Colitis in Adult Japanese Participants (ELEVATE UC 40 JAPAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-308; C5041013 (Other: Alias Study Number)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Etrasimod; APD334; UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily up to 52 weeks
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily up to 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral etrasimod is a safe and effective treatment in adult Japanese participants with moderately to severely active ulcerative colitis (UC). This study is an extension of study APD334-302 (NCT03996369). Participants will continue with the same blinded treatment assigned in Study APD334-302 for a total treatment duration of 52 weeks (12 weeks in Study APD334-302 plus 40 weeks in Study APD334-308).

ELIGIBILITY:
Inclusion Criteria:

Participants with moderately to severely active ulcerative colitis (UC) are eligible to enroll into this study if they fulfill all of the following:

* Must have completed the Week 12 visit of Study APD334-302
* Ability to provide written informed consent or assent (parent or legal guardian must provide consent for a participant < 20 years of age or as required per local regulations who has assented to participate in the study) and to be compliant with the schedule of protocol assessments. Enrollment of participants < 20 years should be conducted only if acceptable according to local laws and regulations.
* Both men and women subjects agree to use a highly effective method of birth control if the possibility of conception exists

Exclusion Criteria:

Participants who meet any of the following exclusion criteria will not be eligible for enrollment into the study:

* If the Investigator considers the participant to be unsuitable for any reason to participate in the study
* Participants requiring partial or total colectomy during the APD334-302 study
* Participants requiring treatment with prohibited concomitant medications

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- Japan (38):
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - Kojunkai Daido Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ishii Eye Clinic, Nagareyama-shi, Chiba
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Takimoto Eye Clinic(OCT), Kasuga-shi, Fukuoka
  - Fakuoka Tokushukai Hospital, Kasuga-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - NHO Mito Medical Center, Higashiibaraki-gun, Ibaraki
  - Matsumoto Eye Clinic, Toride-shi, Ibaraki
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - JA- Kagoshima Koseiren Hospital (PET/DLCO), Kagoshima, Kagoshima-ken
  - Kagoshima Kouseiren Hospital, Kagoshima, Kagoshima-ken
  - Clinical Pathology Laboratory (Diagnostick center), Kagoshima, Kagoshima-ken
  - Jiaikai Idzuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Sameshima Eye Clinic (OCT), Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - National Hospital Organization Kyoto Medical Center, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Mie Prefectural General Medical Center, Yokkaichi-shi, Mie-ken
  - JOHAS Tohoku Rokai Hospital, Sendai, Miyagi
  - JOHAS Tohoku Rosai Hospital, Sendai, Miyagi
  - Sendai City Hospital, Sendai, Miyagi
  - Japan Community Health care Organization Osaka Hospital, Osaka, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Showa General Hospital, Kodaira-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-308

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Comparator: Placebo: Participants received etrasimod matching placebo 1 tablet by mouth, once daily up to 40 weeks in APD334-308
- Experimental: Etrasimod 2 mg: Participants received etrasimod 2 mg tablet by mouth, once daily up to 40 weeks in APD334-308
Period: Treatment
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Started | 14 | 28
Completed | 4 | 18
Not Completed | 10 | 10
Not completed — Disease worsening | 10 | 10
Period: Follow-up
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Started | 14 | 28
Completed | 4 | 18
Not Completed | 10 | 10
Not completed — Lack of Efficacy | 1 | 0
Not completed — Disease worsening | 8 | 10
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg | Total
Number analyzed (Participants) | 14 | 28 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (14.12) | 43.9 (14.29) | 44.0 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 7 | 18 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 28 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 28 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 40 of Study APD334-308
Description: Clinical remission was based on the modified Mayo score (MMS). The MMS is a composite score of 3 assessments consisting of participant-reported symptoms using daily electronic (e)-diary and centrally read endoscopy: stool frequency (SF), rectal bleeding (RB) and endoscopic score (ES). Clinical remission was defined as SF sub-score = 0 (or = 1 with a greater than or equal to [>=] 1-point decrease from Baseline), RB sub-score = 0, and ES less than or equal to (<=) 1 (excluding friability). Each component sub-score ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Week 40 of APD334-308
Population: Full Analysis Set Population (All randomized participants who received at least 1 dose of study intervention). Only those participants with data available at the specified time points were analyzed. "Overall number of participants analyzed" signifies participants evaluable for this outcome measure".
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 7.1 | 25.0
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 17.86, 95% CI 2-sided [-3.10 to 38.82]

2. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 40 of Study APD334-308
Description: Endoscopic improvement was defined as an ES <=1 (excluding friability) at Week 40 of APD334-308 compared with Week 12 of APD334-302. The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease); higher score indicated more severe disease.
Time Frame: Week 40 of APD334-308
Population: Full Analysis Set Population. Only those participants with data available at the specified time points were analyzed. "Overall number of participants analyzed" signifies participants evaluable for this outcome measure".
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 7.1 | 35.7
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 28.57, 95% CI 2-sided [6.28 to 50.86]

3. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Week 40 of Study APD334-308
Description: Symptomatic remission was defined as an SF sub-score = 0 (or = 1 with a >= 1 point decrease from Baseline) and RB sub-score = 0. The SF sub-score ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB sub-score ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicated more severe disease.
Time Frame: Week 40 of APD334-308
Population: Full Analysis Set Population. "Overall number of participants analyzed" signifies participants evaluable for this outcome measure". Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 7.1 | 39.3
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 32.14, 95% CI 2-sided [9.58 to 54.71]

4. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 40 of Study APD334-308
Description: Mucosal healing was defined as an ES <= 1 (excluding friability) with histologic remission measured by a Geboes Index score less than [<] 2.0). The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease). The Geboes score grading system, was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease.
Time Frame: Week 40 of APD334-308
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 7.1 | 28.6
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 21.43, 95% CI 2-sided [-0.07 to 42.92]

5. Secondary Outcome: Percentage of Participants, Who Had Not Been Receiving Corticosteroids for ≥ 12 Weeks, Achieving Clinical Remission at Week 40 of Study APD334-308 Among Participants Receiving Corticosteroids at C5041015 (APD334-302) Study Entry
Description: as for outcome 1
Time Frame: Week 40 of APD334-308
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 7.1 | 25.0
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 17.86, 95% CI 2-sided [-3.10 to 38.82]

6. Secondary Outcome: Percentage of Participants Achieving Sustained Clinical Remission
Description: Clinical remission was based on the modified Mayo score (MMS). The MMS is a composite score of 3 assessments consisting of participant-reported symptoms using daily electronic (e)-diary and centrally read endoscopy: stool frequency (SF), rectal bleeding (RB) and endoscopic score (ES). Clinical remission was defined as SF sub-score = 0 (or = 1 with a greater than or equal to [>=] 1-point decrease from Baseline), RB sub-score = 0, and ES less than or equal to (<=) 1 (excluding friability). Each component sub-score ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease. A subject with sustained clinical remission is defined as someone who achieved clinical remission at both Week 12 of APD334-302 and Week 40 of APD334-308.
Time Frame: Week 40 of APD334-308
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
Number analyzed (Participants) | 14 | 28
Percentage of participants | 0 | 7.1
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: Etrasimod 2 mg; Test type: Other; Risk Difference (RD) = 7.14, 95% CI 2-sided [-2.40 to 16.68]

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) were collected during the 40-week continuous treatment period, followed by a 4-week follow-up period up to Week 44 of C5041013 (APD334-308).
Description: Safety set population included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Placebo Comparator: Placebo | Experimental: Etrasimod 2 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/28
Other Adverse Events (participants affected / at risk) | 8/14 | 16/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: Placebo (N=14) | Experimental: Etrasimod 2 mg (N=28)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: Placebo (N=14) | Experimental: Etrasimod 2 mg (N=28)
Colitis ulcerative (Gastrointestinal disorders) | 1 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 3 (4)
Vaccination site pain (General disorders) | 0 (0) | 2 (3)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 4 (6)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04706793/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT04706793/SAP_002.pdf